CLINICAL TRIAL: NCT01894009
Title: Effect of Foot Manipulation for Relief of Pregnancy Related Pelvic Girdle Pain. A Randomised Clinical Trial in Primary Care
Brief Title: Foot Manipulation for Pregnancy Related Pelvic Girdle Pain
Acronym: PPGP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VGFOUSKB-43121
Record Dates: First submitted 2013-06-20; First posted 2013-07-09 (Estimated); Last update posted 2021-02-05 (Actual); Status verified 2013-07

CONDITIONS: Pregnancy
Keywords: Osteopathic manipulation; Exercise therapy; Pregnancy pelvic girdle pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Foot manipulation (Active Comparator): Asymmetry of the feet was treated by thrusting of the cuboid bone and the subtalar joint was treated with gapping thrust. Mobilisation of the distal tibia-fibula was repeated 10 times. Home training programs in order to maintain the mobility in the joints were given with morning exercises. Four types of exercises were recommended: 1) Foot training with pro-and supination of the feet from dorsal to plantar flexion. 2)"Caterpillar walk". 3) Training the take off of the great toes along a normal walking line and 4) Mobility of lateral malleoli and the talo-crural joint by dorsal flexion of feet while bending the knees.
  Interventions: Procedure: Foot manipulation
- Sham foot manipulation (Sham Comparator): Sham manipulation included downsizing (a massage technique) the section underneath the heel from back forwards with four grips and palpation of the five metatarsal bones with the patient in the supine position on a psoas pillow. Further, light pressure on the Achilles tendon, with the patient standing against a wall with the feet 40 cm off the wall with bent knees on order to simulate the tibio-fibular mobilisation. Home exercises in the mornings to be repeated 8 times.
  Interventions: Procedure: Sham foot manipulation

INTERVENTIONS:
Procedure: Foot manipulation — The subtalar joint was treated with gapping thrust with patient lying on the contra-lateral side. Mobilisation of the distal tibia-fibula was performed with the patient squatting and was repeated 10 times. Home training programs in order to maintain the mobility in the joints were given.
  Arms: Foot manipulation
Procedure: Sham foot manipulation — Sham manipulation included downsizing (a massage technique) the section underneath the heel from back forwards with four grips and palpation of the five metatarsal bones. Sham manipulations were repeated 10 times. This group was also recommended home exercises in the mornings.
  Arms: Sham foot manipulation

SUMMARY:
Background: Asymmetrical foot posture influences the pelvic girdle stability and might give pain in the pelvic region. The objective was to investigate if foot manipulation to correct foot asymmetry can relieve pregnancy related pelvic girdle pain (PPGP) and shorten sick leave periods.

Design: Randomized single blinded (patients and evaluators) clinical trial comparing foot with sham manipulation at 6 weekly treatment sessions.

Setting: Five physiotherapy out-patient clinics (10 physiotherapists) in Skaraborg Primary Care, Sweden.

DETAILED DESCRIPTION:
The study was performed at the physiotherapy clinics at five Health Care Centres in Skaraborg from September 2009 to August 2011. Women with suspected PPGP were referred by midwifes or physicians or contacted the physiotherapists directly. Inclusion criteria were Swedish-speaking women in gestational weeks 12-31 with PPGP determined by specific provocation tests, including the 4P test (posterior pelvic pain provocation test), Patrick's test, ASLR (active straight leg raise test), modified Trendelenburg test and palpation of symphysis pubis. Women with twin pregnancies, lumbar pain, rheumatic or other serious disease were excluded as well as non-Swedish-speaking woman and those who had had foot manipulation earlier. The feet were inspected in standing position to estimate whether they were straight, rotated outwards or inwards and if the load was flat, pronated or supinated. Movement in the subtalar joints was investigated as well as elasticity of the tarsal bones and the lateral malleoli. All women that were included had asymmetric position of one or both feet.

Study procedure Patients were randomized to either foot or sham manipulation using sealed envelopes (n=150; 75 for each treatment). The envelopes were administered and mixed centrally and depending on size the physiotherapy clinic were assigned an appropriate number of envelopes. Ten physiotherapists participated pair-wise in the treatments, one treated the patient (physiotherapist unblinded, patient blinded), and the other made the evaluation (double blinded). All patients got the same information about PPGP and 6 visits once a week during 6 weeks, and follow-up visits one week after end of treatment and three months after delivery. All patients were encouraged not to talk to other pregnant women or to the evaluators about details of their treatment.

Data were registered in protocols separated from the medical records, not accessible for the evaluators, and included group assignment, results of diagnostic tests, Vorlauf tests and Visual Analogue Scales (VAS). The blinded evaluator administered the follow-up three months after delivery.

ELIGIBILITY:
Inclusion Criteria:

Women with suspected PPGP were referred by midwifes or physicians or contacted the physiotherapists directly.

Inclusion criteria:

* Swedish-speaking women in gestational weeks 12-31
* Pregnancy Related Pelvic Girdle Pain (PPGP) determined by provocation tests (4P test, posterior pelvic pain provocation test; Patrick's test, ASLR (active straight leg raise test), modified Trendelenburg test and pain on palpation of symphysis pubis

Exclusion Criteria:

Women with:

* twin pregnancies
* lumbar pain
* rheumatic or other serious disease
* non-Swedish-speaking woman
* those who had had experinced foot manipulation earlier

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Difference in Pregnancy related pelvic girdle pain and Vorlauf test outcome | Before and after treatment at assessments during 6 weeks and three months after childbirth.
  Pain reduction:
  Pain in pelvic girdle,(pain in pelvis, sacroiliac joint (SIJ) and symphysis)during 6 weeks after start of treatment and 3 months after childbirth using VAS a diary with VAS graded from 0 to 100 rating their pain each morning and evening.
  Vorlauf test:
  Both posterior superior iliac spines (PSIS) were identified with the patient sitting by a grip underneath the lower edge of the spines. The grip was maintained as the patient rose and the levels of the PSIS were noted. If the levels differed (positive Vorlauf test), the lowest was compensated with a plate measuring 2-5 mm under the corresponding foot after which, the patient bent forward to evaluate Vorlauf. Thwew tests were performed by a physiotherapist blinded to the kind of treatment the woman was exposed to. An asymmetric movement of PSIS indicated a locking of the sacroiliac joint.

SECONDARY OUTCOMES:
Change in number of days of Sick leave | Before and after treatment at assessments during 6 weeks.
  Sick leave:
  During 6 weeks after start of treatment and 3 months after childbirth using a diary in which they indicated whether they were on sick leave 25%, 50%, 75% or 100% of full time. Net days of sick leave were calculated as the number of days multiplied with the degree of sick leave.

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Melkersson, Physiother, Principal Investigator — R&D Centre, Skaraborg Primary Care, Skövde, Sweden
Locations (1):
- Närhälsan Tibro Rehabmottagningen, Centrumgatan 11-17, Tibro, Sweden